CLINICAL TRIAL: NCT06173193
Title: Effects of a Multicomponent Exercise Regimen on Subchondral Bone, Cartilage, and Inflammation Markers in Postmenopausal Women with Knee Osteoarthritis: a Randomized Controlled Study
Brief Title: Effects of Multicomponent Exercise on Subchondral Bone and Cartilage in Postmenopausal Women with Knee Osteoarthritis
Acronym: LuRu2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: University of Oulu (Other); Wellbeing Services County of Central Finland (Unknown); UKK Institute (Other); Research Council of Finland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21000057531; 351483 (Other Grant/Funding Number: Academy of Finland)
Record Dates: First submitted 2023-10-31; First posted 2023-12-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Exercise; Subchondral bone; Cartilage; Randomized controlled trial; Postmenopausal women; Osteoarthritis; Physiotherapy; Joint Diseases; Musculoskeletal Diseases; Physical functioning
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Osteoarthritis; Joint Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- multicomponent exercise group (Experimental): 8 months of multicomponent exercise (3 sessions/week).
  Interventions: Behavioral: Multicomponent exercise regimen
- Reference group (Active Comparator): 8 months of standard rehabilitative care based home exercises.
  Interventions: Behavioral: Standard rehabilitative management

INTERVENTIONS:
Behavioral: Multicomponent exercise regimen — A multicomponent exercise regimen applied is comprised of the step-aerobic and resistance training programs alternating every two weeks. The trainees participate in supervised training sessions 3 times a week for 8 months. Each session will include a 10-minutes warm-up, 30-minutes of effective training part and a 10-minutes period for cooling down.
  Step-aerobic: The program includes accelerating and decelerating through forwards and sideways movements with stops and turns to music. The degree of difficulty of movements and steps as well as training intensity will be gradually increased by increasing the height of the step benches.
  Resistance training: The participants will undergo a progressive resistance training program. Resistance training will emphasize training of following muscle groups: Quadriceps and hamstrings, hip abductors, adductors and extensors, and calf muscles. In addition to lower limb exercises, trunk and upper body exercises will be applied at intervals.
  Arms: multicomponent exercise group
Behavioral: Standard rehabilitative management — The treatments that will be provided to the members of a reference group represent the standard rehabilitative management for knee OA patients. The home exercises focus on functional exercises maintaining lower extremity flexibility and muscle function. The home exercises are instructed to be carried out three times a week, each work-out lasting 30 minutes.
  Arms: Reference group

SUMMARY:
Today, osteoarthritis (OA) is considered a whole-organ disease that is amenable to prevention and treatment in the early stages. Information on the articular cartilage and subchondral bone responses to exercise may help to develop safe and feasible exercise programs which can potentially improve cartilage and bone properties. Therefore, the goal of this study is to produce the knowledge needed to understand what effects multicomponent exercise regimen have on subchondral bone and articular cartilage of the knee joint in postmenopausal women with knee OA.

Participants will be randomized into either:

1. Intervention group, which conducts multicomponent exercise regimen including alternating step-aerobic and resistance training.
2. Reference group, which represents the standard rehabilitative management for knee OA patients with home exercises.

Researchers will compare intervention and reference groups to see if subchondral bone morphology and properties and cartilage biochemical alterations differ between the groups at the end of the 8-month intervention and 12-month follow-up period.

DETAILED DESCRIPTION:
The study is an 8-month, randomized controlled intervention study with 12-month follow-up in volunteer postmenopausal (55-75-year-old) women with mild radiographic knee OA according to the Kellgren-Lawrence classification (grade 1-2). The participants will be randomly assigned into the subgroups. The study will be conducted in two phases.

8-month multicomponent exercise regimen will be carried out gradually and progressively three times a week by experienced and recently trained exercise instructors. The instructors will keep an attendance and an adverse event record for each of the intervention group's participants. The home exercises carried out three times a week by the reference group represent the standard rehabilitative management for knee OA patients.

In addition to the above-mentioned treatments, all participants will receive instructions to use paracetamol on an as-needed basis. Participants will be called to end-point measurements at 8 months after baseline and follow-up measurements at 20 months after baseline.

The overall goal of this study is to produce the knowledge needed to understand what effects multicomponent exercise regimen have on subchondral bone and articular cartilage of the knee joint in postmenopausal women with knee OA. In addition, the aim is to develop means to improve functional competence as well as to prevent physical disability among women suffering from knee OA. Specifically, the objectives are to investigate the effects of joint loading exercise regimen on knee joint subchondral bone morphology and properties, and cartilage biochemical alterations and their 12 month maintenance in women with knee OA. Also, training effects on molecular biomarkers related to OA and inflammation, bone traits, physical function, performance, body composition, and clinically important symptoms will be examined.

ELIGIBILITY:
Inclusion Criteria:

* voluntary women 55-75 years of age.
* no history of any illness for which exercise is contraindicated or that would limit participation in the exercise program.
* knee pain during the last 12 months.
* willingness and voluntarily signed informed consent to undergo testing and intervention procedures with all of its aspects.
* weight-bearing knee x-rays show radiographic Kellgren-Lawrence grade 1-2 OA in one or both tibiofemoral joints.

Exclusion Criteria:

* body-mass index over 35 kg/m2.
* knee instability or trauma that would jeopardize the training.
* inflammatory joint disease.
* intra-articular steroid injections in the preceding 12 months in the knee.

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Tibiofemoral articular cartilage's glycosaminoglycan content | Baseline, 8 months, 20 months
  Assessed by quantitative Magnetic Resonance Imaging (qMRI) techniques at 3Tesla MR-system. Rotating frame of reference contrast adiabatic T1rho (ms) will be measured.
Tibiofemoral articular cartilage's collagen content and orientation | Baseline, 8 months, 20 months
  T2 maps (ms) will be assessed by qMRI techniques at 3Tesla MR-system. In addition, some clinical MRI series will be conducted.
Tibiofemoral articular cartilage thickness (mm) | Baseline, 8 months, 20 months
  Assessed by 3D-texture analysis.
Tibiofemoral articular cartilage volume (mm^3) | Baseline, 8 months, 20 months
  Assessed by 3D-texture analysis.
Tibiofemoral subchondral bone mineral density (g/cm^3) | Baseline, 8 months, 20 months
  Assessed by high-resolution cone beam computed tomography (CBCT).
Tibiofemoral subchondral bone mineral content (g) | Baseline, 8 months, 20 months
  Assessed by high-resolution CBCT.
Tibiofemoral joint space narrowing (mm) | Baseline, 8 months, 20 months
  Assessed by high-resolution CBCT.

SECONDARY OUTCOMES:
Bone mineral content (BMC, g) of the femoral neck | Baseline, 8 months, 20 months
  Assessed by Dual-energy X-ray absorptiometry (DXA).
Areal bone mineral density (aBMD, g/cm^2) of the femoral neck | Baseline, 8 months, 20 months
  Assessed by DXA.
Cortical thickness (mm) of the femoral neck | Baseline, 8 months, 20 months
  Assessed by Advanced Hip Analysis software.
Femoral neck width (mm) | Baseline, 8 months, 20 months
  Assessed by Advanced Hip Analysis software.
Cross-sectional area (cm^2) of the femoral neck | Baseline, 8 months, 20 months
  Assessed by Advanced Hip Analysis software.
Cross-sectional moment of inertia (cm^4) of the femoral neck | Baseline, 8 months, 20 months
  Assessed by Advanced Hip Analysis software.
Section modulus (cm^3) of the femoral neck | Baseline, 8 months, 20 months
  Assessed by Advanced Hip Analysis software.
Total body fat percentage (%) | Baseline, 8 months, 20 months
  Assessed by DXA.
Fat Free Mass Index (FFMI, kg/m^2) | Baseline, 8 months, 20 months
  Assessed by DXA.
Clinically important OA-symptoms and physical function | Baseline, 8 months, 20 months
  Assessed by Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire (Score 0-100). Higher scores represent better outcomes.
Health-related quality of life | Baseline, 8 months, 20 months
  Assessed by RAND 36-Item Health Survey questionnaire (Scores 0-100 on different domains). Higher scores represent a more favorable health state.
Work disablement | Baseline, 8 months, 20 months
  Assessed by short form of Örebro musculoskeletal pain screening questionnaire (Score 1-100). Higher scores estimate increased risk for future work disability.
Self-rated physical activity | IPAQ: Baseline, 8 months, 20 months. Physical activity diary: through the 8-month study intervention in the control group
  Assessed by International Physical Activity Questionnaire (IPAQ, Metabolic equivalent task (MET) -minutes). Also, physical activity diary (MET-minutes) will be filled by the control group through the 8-month study intervention.
Objective daily physical activity | See above
  Assessed by a tri-axial accelerometer (minutes & MET-hours), worn 24 hours a day. A tri-axial accelerometer will be used through the 8-month study intervention in the intervention group and periods of 7 consecutive days every two months during the 8-month study intervention in the control group. During the 12-month follow-up, all the participants will be measured every four months for seven consecutive days.
Quantity of painkillers consumed | Through the 8-month study intervention
  Assessed by diary.
Systemic inflammation markers | Baseline, 8 months, 20 months
  High sensitivity C-reactive protein and serum cytokines including interleukin-6 and tumor-necrosis factor alpha will be assessed from blood.
Metabolic profile | Baseline, 8 months, 20 months
  Circulating metabolomes including resistin, leptin, adiponectin, lipids, lipoproteins, and metabolites will be assessed from blood.
Cardiorespiratory fitness | Baseline, 8 months, 20 months
  Assessed by UKK 2km walk test (minutes and seconds).
Knee extension and flexion maximal isometric muscle strength | Baseline, 8 months, 20 months
  Assessed by an adjustable dynamometer chair (Newtons).
Static balance | Baseline, 8 months, 20 months
  Assessed by a single leg stance test (seconds).
30 second chair-stand test (seconds) | Baseline, 8 months, 20 months
Timed up and go (TUG) (seconds) | Baseline, 8 months, 20 months
40m Fast-paced walk test (seconds) | Baseline, 8 months, 20 months
Stair climb test (seconds) | Baseline, 8 months, 20 months
Walking biomechanics | Baseline, 8 months, 20 months
  Lower body's segmental acceleration (m/s^2) in 40m Fast-paced walk test, Stair climb test, and 2-minute walk at the subject's preferred pace will be assessed by Inertial Measurement Unit (IMU).

CONTACTS AND LOCATIONS:
Overall Officials: Ari Heinonen, Prof., emeritus, Principal Investigator — University of Jyvaskyla
Locations (1):
- University of Jyväskylä, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No
IPD cannot be anonymized and will thus remain restricted due to personal data protection. The basic project-level discovery metadata of the dataset(s) will be made openly available in the University's repository with a DOI for permanent findability and accessibility whenever the metadata are sufficiently complete to be published.

REFERENCES:
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Derived] Konola VM, Parkkari J, Multanen J, Nikander R, Rantalainen T, Vesanto J, Pekkala S, Kalaja M, Ihalainen JK, Waller B, Munukka M, Sievanen H, Nevalainen M, Kautiainen H, Casula V, Paloneva J, Vasankari T, Peuna A, Saarakkala S, Nieminen MT, Heinonen A. Effects of a multicomponent exercise regimen on subchondral bone and cartilage in postmenopausal women with knee osteoarthritis: protocol for a randomized controlled trial. Trials. 2025 Jun 23;26(1):222. doi: 10.1186/s13063-025-08928-1. PMID 40551179